CLINICAL TRIAL: NCT02797626
Title: Phase II Single-arm Trial to Evaluate Progression Free Survival With Primary Retroperitoneal Lymph-node Dissection (pRPLND) Only in Patients With Seminomatous Testicular Germ Cell Tumors With Clinical Stage IIA/B (PRIMETEST)
Brief Title: Trial to Evaluate Progression Free Survival With Primary Retroperitoneal Lymph-node Dissection (pRPLND) Only in Patients With Seminomatous Testicular Germ Cell Tumors With Clinical Stage IIA/B (PRIMETEST)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015053664
Record Dates: First submitted 2016-06-08; First posted 2016-06-13 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Stage II A/B Seminomatous Germ Cell Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Primary RPNLD (Other)
  Interventions: Procedure: Primary retroperitoneal lymph-node dissection (pRPLND)

INTERVENTIONS:
Procedure: Primary retroperitoneal lymph-node dissection (pRPLND) — Open or laparoscopic robotic-assisted nerve-sparing retroperitoneal lymph node dissection (modified template RPLND, if possible ipsilateral nerve-sparing)

SUMMARY:
Primary objective:

to evaluate progression-free survival in patients with clinical stage II A/B seminomatous germ cell tumor undergoing primary retroperitoneal lymph node dissection (RPLND) without adjuvant treatment

Secondary objectives:

* overall survival
* perioperative complications (Clavien-Dindo score)
* quality of life (EORTC QLQ C30, EORTC QLQ TC26)
* long term sequelae
* rate of retrograde ejaculation

DETAILED DESCRIPTION:
Standard treatment of patients with clinical stage IIA seminoma (isolated retroperitoneal lymph nodes up to 2 cm) is radiotherapy (30Gy) and for clinical stage IIB (isolated retroperitoneal lymph nodes 2-5 cm) is radiotherapy (36Gy, extended iliac field). Alternatively, 3 courses of BEP are equal (1,2,3,4). According to the EAU guidelines 3 cycles of BEP can be substituted for 4 x PE in patients with contraindications for bleomycin. Radiotherapy as well as chemotherapy has several side effects: multiple studies show significant long term toxicity after cisplatin chemotherapy such as cardiotoxicity or nephrotoxicity (5,6,7,8, 9). Patients after radiotherapy show a significant increased rate of secondary malignancies during long term follow-up (relative risk between 1.3 and 1.4) (13, 14).

There are no reliable data on recurrences of patients with seminoma in CS II who have undergone surgery only. After the publication of Warszawski et al in 1997 primary RPLND in seminoma has not been performed on a routine basis (10). However, seminoma metastasis follows the same anatomical principles as non-seminoma and is primarily lymphatic. In clinical stage I high risk seminoma patients the overall recurrence rate without adjuvant therapy is ~ 30%, in CS IIB patients after radiotherapy at around 18%, respectively (11,12). If seminoma stage II patients could achieve a less than 10% recurrence rate after surgery, surveillance as well as a single course adjuvant chemotherapy would again be justified. The overall burden of standard treatment with 3 or 4 courses of chemotherapy could thereby considerably reduced. With a recurrence rate of > 30% (exceeding the upper border of the confidence interval) every third patient would require surgery and chemotherapy and the overall treatment burden would not justify this approach.

Thus, the hypothesis of this trial is currently an overtreatment of patients with low volume metastasis either initially diagnosed or as recurrence with 3 courses BEP chemotherapy as recommended standard treatment in most of these patients. In addition, surgical techniques have evolved and laparoscopic robot-assisted RPLND seems possible in unilateral low stage disease.

In order to clarify the role of primary RPLND in this patient cohort, the progression-free survival has to be explored in a single arm non-randomized trial. Only if the recurrence rate does not exceed the published figures further adjuvant treatment is justified. In a subsequent trial patients may then be selected based on prognostic parameters to receive surveillance after primary RPLND only or to be treated by 1 course of BEP in cases of higher relapse figures. Therefore, this trial may serve as first step to improve the overall treatment burden in patients with clinical stage II disease.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed seminomatous testicular germ cell tumor
* inguinal, paraaortic or retroperitoneal lymph nodes classified as local or regional unilateral lymph node metastasis by contrast CT or MRI
* maximum dimensions of lymph node metastasis: single mass of max. 5.0 cm in transverse CT diameter multiple metastases in a unilateral field with single max. diameter of 5.0 cm (UICC IIB)

patients with serum tumour marker elevation at the time of CT staging are eligible if the elevated human chorionic gonadotropin (hCG) directly before RPLND does not exceed 5 IU/L

* patients qualify for this trial with following scenarios

  1. initial diagnosis of UICC clinical stage IIA/IIB disease
  2. recurrence after surveillance for clinical stage I
  3. recurrence after adjuvant treatment of clinical stage I seminoma with 1 x carboplatin AUC7
* curative treatment is intended
* patient´s age above 18 years
* able to communicate well with the investigator, to understand and comply with the requirements of the study, to understand and sign the written informed consent.

Exclusion Criteria:

* non-seminomatous germ cell tumors
* germ cell tumor-related AFP elevation suspicious of non-seminoma
* metastatic lymph node mass with greatest dimension >5 cm (CS IIC)
* other metastasis (CS III)
* patients with prior scrotal or retroperitoneal surgery due to other diseases than germ cell cancer
* patient underwent chemotherapy other than adjuvant Carboplatin monotherapy
* patient underwent radiotherapy of the retroperitoneum
* patient in reduced general condition or with live threatening disease
* patient has a psychiatric disease
* patient does not have sufficient knowledge of German language

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06; Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Albers, M.D., PhD, Principal Investigator — Department of Urology, Heinrich Heine University, Duesseldorf, Germany; Achim Lusch, M.D., Principal Investigator — Department of Urology, Heinrich Heine University, Duesseldorf, Germany
Locations (1):
- Departement of Urology, Heinrich Heine University Duesseldorf, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided